CLINICAL TRIAL: NCT04640623
Title: Phase 2b Clinical Study Evaluating Efficacy and Safety of TAR-200 in Combination With Cetrelimab, TAR-200 Alone, or Cetrelimab Alone in Participants With High-Risk Non-Muscle Invasive Bladder Cancer (NMIBC) Unresponsive to Intravesical Bacillus Calmette-Guérin (BCG) Who Are Ineligible for or Elected Not to Undergo Radical Cystectomy
Brief Title: A Study of TAR-200 in Combination With Cetrelimab, TAR-200 Alone, or Cetrelimab Alone in Participants With Non-Muscle Invasive Bladder Cancer (NMIBC) Unresponsive to Intravesical Bacillus Calmette-Guérin Who Are Ineligible for or Elected Not to Undergo Radical Cystectomy
Acronym: SunRISe-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108921; 17000139BLC2001 (Other: Janssen Research & Development, LLC); 2020-002646-16 (EudraCT Number); 2023-506146-23-00 (Registry Identifier: EUCT number)
Expanded Access: NCT06877676 (Approved for marketing)
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: TAR-200 and Cetrelimab (Experimental): TAR-200 is placed into the bladder through a urinary placement catheter in participants with carcinoma in situ (CIS), with or without papillary disease, on Day 0 and will be dosed every 3 weeks (Q3W) for up to the first 24 weeks (6 months), then every 12 weeks through Week 99 (Year 2). In addition, Cetrelimab will be dosed Q3W through Week 78 (18 months).
  Interventions: Drug: TAR-200; Biological: Cetrelimab
- Cohort 2: TAR-200 (Experimental): TAR-200 is placed into the bladder through a urinary placement catheter in participants with CIS, with or without papillary disease, on Day 0 and will be dosed Q3W for up to the first 24 weeks (6 months), then every 12 weeks through Week 99 (Year 2).
  Interventions: Drug: TAR-200
- Cohort 3: Cetrelimab (Experimental): Participants with CIS, with or without papillary disease, will receive Cetrelimab which will be dosed Q3W through Week 78 (18 months).
  Interventions: Biological: Cetrelimab
- Cohort 4: TAR-200 (Participants with Papillary Disease only) (Experimental): TAR-200 is placed into the bladder through a urinary placement catheter in participants with papillary disease only, on Day 0 and will be dosed Q3W for up to the first 24 weeks (6 months), then every 12 weeks through Week 99 (Year 2).
  Interventions: Drug: TAR-200

INTERVENTIONS:
Drug: TAR-200 — TAR-200 will be administered transuretherally.
  Other Names: JNJ-17000139; Gemcitabine-Releasing Intravesical System
  Arms: Cohort 1: TAR-200 and Cetrelimab; Cohort 2: TAR-200; Cohort 4: TAR-200 (Participants with Papillary Disease only)
Biological: Cetrelimab — Cetrelimab will be administered.
  Other Names: JNJ-63723283
  Arms: Cohort 1: TAR-200 and Cetrelimab; Cohort 3: Cetrelimab

SUMMARY:
The purpose of this study is to evaluate the overall complete response (CR) rate in participants treated with TAR-200 in combination with cetrelimab (Cohort 1), or TAR-200 alone (Cohort 2), or cetrelimab alone (Cohort 3) with Carcinoma in Situ (CIS), with or without concomitant high-grade Ta or T1 papillary disease; and disease-free survival (DFS) in participants treated with TAR-200 alone with papillary disease only (Cohort 4).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of persistent or recurrent high-risk non-muscle invasive bladder cancer (HR-NMIBC), (carcinoma in situ [CIS] or tumor in situ [Tis]), with or without papillary disease (T1, high-grade Ta) or papillary disease only (high-grade Ta or any T1 and absence of CIS), within 12 months of completion of the last dose of Bacillus Calmette-Guerin (BCG) therapy, in participants who have received adequate BCG. Mixed histology tumors are allowed if urothelial differentiation (transitional cell histology) is predominant. However, the presence of neuroendocrine, micropapillary, signet ring cell, plasmacytoid, or sarcomatoid features will make a participant ineligible. For participants with lamina propria invasion (T1) on the screening biopsy/ transurethral resection of bladder tumor (TURBT), muscularis propria must be present in order to rule out Muscle Invasive Bladder Cancer (MIBC)
* All visible papillary disease must be fully resected (absent) prior to randomization (residual CIS is acceptable for participants eligible for Cohorts 1, 2, and 3 only) and documented in the electronic case report form (eCRF) at screening cystoscopy. For participants with papillary disease only (Cohort 4), local urine cytology at screening must be negative or atypical (for High-Grade Urothelial Carcinoma [HGUC])
* Participants must be ineligible for or have elected not to undergo radical cystectomy
* BCG-unresponsive high-risk NMIBC after treatment with adequate BCG therapy defined as a minimum of 5 of 6 full doses of an induction course (adequate induction) plus 2 of 3 doses of a maintenance course, or at least 2 of 6 doses of a second induction course
* Eastern Cooperative Oncology Group (ECOG) performance status Grade 0, 1, or 2

Exclusion Criteria:

* Presence or history of histologically confirmed, muscle-invasive, locally advanced, nonresectable, or metastatic urothelial carcinoma (that is, T2, T3, T4, and/or Stage IV)
* Must not have had urothelial carcinoma or histological variant at any site outside of the urinary bladder. Ta/T1/CIS of the upper urinary tract (including renal pelvis and ureter) is allowable if treated with complete nephroureterectomy more than 24 months prior to randomization
* Received a live virus vaccine within 30 days prior to the initiation of study treatment. Inactivated (non-live or non-replicating) vaccines approved or authorized for emergency use (for example, COVID-19) by local health authorities are allowed
* Active hepatitis B or C infection (for example, participants with history of hepatitis C infection but undetectable hepatitis C virus polymerase chain reaction (PCR) test and participants with history of hepatitis B infection with positive hepatitis B surface antigen (HBsAg) antibody and undetectable PCR are allowed)
* Prior therapy with an anti-programmed-cell death 1 (PD-1), anti-PD-ligand 2 (L2) agent, or with an agent directed to another co-inhibitory T-cell receptor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1, 2, and 3: Overall Complete Response (CR) Rate | Up to 5 years
  Overall CR rate is defined as the percentage of participants achieving a CR at any time post-treatment. It will be measured by determining the percentage of participants without presence of high-grade disease using results from cystoscopy and centrally read urine cytology at any time point.
Cohort 4: Disease-free Survival (DFS) | Up to 5 years
  DFS will be measured as the time from the date of first dose of study treatment to either the time of the first recurrence of high-risk disease, progression, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Cohort 1, 2, and 3: Duration of Response (DOR) | Up to 5 years
  DOR is defined from the date of first CR achieved to the date of first evidence of recurrence or progression or death (whichever is earlier) for participants who achieve a CR.
Overall Survival (OS) | Up to 5 years
  OS, defined as the time from the date of first dose of study treatment to death; if a participant has not died at the time of analysis, the participant will be censored at the date last known alive.
Cohort 1, 2, and 4: Concentrations of Gemcitabine and 2',2' difluorodeoxyuridine (dFdU) in Urine and Plasma | Up to Week 21
  Concentrations of gemcitabine and its metabolite dFdU in urine and plasma will be assessed.
Cohort 1 and 3: Serum Concentration of Anti-cetrelimab Antibodies | Predose, up to 3 years
  Serum concentration of anti-cetrelimab antibodies will be assessed using a validated immunoassay for anti-drug antibody (ADA) analysis.
Number of Participants with Anti-cetrelimab Antibodies | Predose, up to 3 years
  Number of participants with anti-cetrelimab antibodies will be reported.
Change from Baseline in European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire (EORTC QLQ) -C30 Scores | Baseline, up to 3 years and 4 months
  EORTC QLQ-C30 is a core 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies. It incorporates 5 functional scales (physical, role, cognitive, emotional, and social functioning), 3 symptom scales (fatigue, pain, and nausea or vomiting), and a global health status or HRQoL scale. Ratings for each item range from 1 (not at all) to 4 (very much).
Change from Baseline in EORTC QLQ- Non-Muscle-Invasive Bladder Cancer (NMIBC) 24 Scores | Baseline, up to 3 years and 4 months
  EORTC QLQ-NMIBC24 is a 24-item questionnaire for evaluating the HRQoL of participants with superficial (non-muscle-invasive) bladder cancer. The questionnaire is designed to supplement the QLQ-C30 and incorporates 6 multi-item scales and 5 single items. Ratings for each item range from 1 (not at all) to 4 (very much).
Number of Participants with Adverse Events (AEs) by Severity Grades | Up to 5 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity grades ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (143):
- United States (22):
  - Del Sol Research Management, LLC, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Genesis Healthcare Partners - Genesis Research Greater Los Angeles, Sherman Oaks, California
  - The Urology Center of Colorado, Denver, Colorado
  - Foothills Urology - Golden Off, Golden, Colorado
  - DuPage Medical Group, Lisle, Illinois
  - Urology of Indiana, Greenwood, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - Michigan Institute of Urology, Troy, Michigan
  - NYU Langone Health, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Associated Medical Professionals, Syracuse, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Urology Associates, PC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Spokane Urology, Spokane, Washington
- Australia (3):
  - Flinders Medical Centre, Bedford Park
  - Eastern Health Research, Box Hill
  - Macquarie University Hospital, Sydney
- Belgium (7):
  - Algemeen Ziekenhuis Sint-Jan, Assebroek
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - Hopital Erasme, Brussels
  - Algemeen ziekenhuis Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Algemeen Ziekenhuis Delta, Roeselare
  - AZ Nikolaas, Sint-Niklaas
- Canada (5):
  - Exdeo Clinical Research Inc, Abbotsford, British Columbia
  - William Osler Health System, Brampton, Ontario
  - Princess Margaret Hospital- UHN, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Universite de Sherbrooke, Sherbrooke, Quebec
- France (20):
  - Hopital Pellegrin CHU Bordeaux, Bordeaux
  - Polyclinique Bordeaux Nord Acquitaine, Bordeaux
  - CHU Grenoble, Grenoble
  - Clinique Sainte Marguerite, Hyères
  - Polyclinique de Limoges - Francois Chenieux, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre de Cancerologie du Grand Montpellier, Montpellier
  - CHU Nimes, Nîmes
  - Hopital Saint Louis, Paris
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Clinical La Croix Du Sud - Ramsay Santé, Quint-Fonsegrives
  - Hopital Pontchaillou, Rennes
  - CHP Saint Gregoire, Saint-Grégoire
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
  - Hopital Foch, Suresnes
  - Hopital Rangueil, Toulouse
- Germany (9):
  - Urologische Partnerschaft Koln UPK, Cologne
  - Urologicum Duisburg, Duisburg
  - Klinikum Herne - Urologie, Herne
  - Matthias Schulze - Germany, Markkleeberg
  - Urologie Neandertal Praxis Mettmann, Mettmann
  - Universitatsklinikum Munster, Münster
  - Schön Klinik Nürnberg Fürth, Nuremberg
  - Studienpraxis Urologie Nürtingen - Germany, Nürtingen
  - Urologische Praxis am Wasserturm - Germany, Würselen
- Greece (6):
  - Metropolitan General A E, Cholargós
  - Athens Medical Center, Marousi
  - Bioclinic - Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki G. Gennimatas, Thessaloniki
  - Euromedica General Clinic, Thessaloniki
  - Papageorgiou General Hospital Of Thessaloniki, Thessaloniki
- Italy (10):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Sant Andrea, Roma
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale San Bortolo, Vicenza
- Japan (11):
  - Aso Co.,Ltd Iizuka Hospital, Iizuka
  - St Marianna University Hospital, Kanagawa
  - Nara Medical University Hospital, Kashihara-shi
  - Kimitsu Chuo Hospital, Kisarazu-shi
  - Nagasaki University Hospital, Nagasaki
  - JOHAS Osaka Rosai Hospital, Osaka
  - Toranomon Hospital, Tokyo
  - Toyama University Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - University of Tsukuba Hospital, Tsukuba
  - Yokohama City University Medical Center, Yokohama
- Netherlands (4):
  - Antoni van Leeuwenhoek, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - The Julius Center - Utrecht Science Park - Stratenum, Utrecht
- Portugal (9):
  - Hospital Garcia de Orta, Almada
  - Uls Regiao Aveiro - Hosp. Infante D. Pedro, Aveiro
  - Uls Alto Ave - Hosp. Sra. Da Oliveira Guimaraes, Guimarães
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Fund. Champalimaud, Lisbon
  - Uls Loures Odivelas - Hosp. Loures, Loures
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, Porto
  - Centro Hospitalar de Vila Nova de Gaia Espinho E P E, Vila Nova de Gaia
  - Centro Hospitalar de Trás os Montes e Alto-Douro, Vila Real
- Russia (9):
  - Hertzen Oncology Research Institute, Moscow
  - Privolzhsky District Medical Centre, Nizhny Novgorod
  - Avicenna Medical Center, Novosibirsk
  - A. Tsyb Medical Radiological Research Center, Obninsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - Ultrasound Clinic 4D, Pyatigorsk
  - Saratov State Medical University, Saratov
  - Multifunctional clinical medical center 'Medical city', Tyumen
  - Bashkir State Medical University, Ufa
- South Korea (10):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (13):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Fund. Puigvert, Barcelona
  - Hosp. Puerta Del Mar, Cadiz
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Instituto Valenciano de Oncologia, Valencia
- Ukraine (3):
  - Chernihivskyi oblasnyi onkolohichnyi dyspanser, Chernihiv
  - Asklepion LLC, Kiev
  - Sumy Regional Clinical Oncology Centre, Sumy
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Daneshmand S, Van der Heijden MS, Jacob JM, Guerrero-Ramos F, Bogemann M, Simone G, Pieczonka CM, Casco NC, Zainfeld D, Spiegelhalder P, Xylinas E, Cahn D, Lotan Y, Murray KS, Kawahara T, Stromberg K, Martin J, Shukla A, Cutie CJ, Bertzos K, Hampras S, Sweiti H, Necchi A; SunRISe-1 Study. TAR-200 for Bacillus Calmette-Guerin-Unresponsive High-Risk Non-Muscle-Invasive Bladder Cancer: Results From the Phase IIb SunRISe-1 Study. J Clin Oncol. 2025 Nov 20;43(33):3578-3588. doi: 10.1200/JCO-25-01651. Epub 2025 Jul 30. PMID 40737582